CLINICAL TRIAL: NCT06092164
Title: Visual Outcomes of Different Types of Functional Intraocular Lenses in Cataract Patients
Brief Title: Visual Outcomes of Functional Intraocular Lenses in Cataracts
Status: Not yet recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jin Yang, Professor, Eye & ENT Hospital of Fudan University
Other Study IDs: IOL Outcomes in cataracts
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cataract; Visual Quality
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, multi-center, randomized comparative study. The purpose of the study is to evaluate and compare the objective and subjective visual outcomes of different types of functional intraocular lenses (IOLs) in patients.

DETAILED DESCRIPTION:
Analyzing the subjective and objective visual outcomes and related factors following the implantation of various types of intraocular lenses（bifocal, trifocal, extended depth of focus (EDOF), and astigmatism-correcting intraocular lenses), exploring the advantages, disadvantages, and suitable patient populations for different types of intraocular lenses, analyzing the factors affecting postoperative visual quality, and providing guidance to better assist patients with diverse needs in clinical settings, aiming to offer multidimensional postoperative visual quality."

ELIGIBILITY:
Inclusion Criteria:

* cataract
* age > 18 years

Exclusion Criteria:

* amblyopia; previous ocular surgery;
* ocular pathologies such as diabetic retinopathy, macular degeneration, glaucoma with field defects;
* requirements for further ocular surgery (other than Nd:YAG capsulotomy) or retinal laser treatments during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Catarct
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
uncorrected distance visual acuity (UDVA) | one year
  uncorrected visual acuity at 5 m
best corrected distance visual acuity (BCVA) | one year
  corrected visual acuity at 5 m
uncorrected near visual acuity (UNVA) | one year
  uncorrected visual acuity at 40 cm
uncorrected intermediate visual acuity (UIVA) | one year
  uncorrected visual acuity at 60 cm

SECONDARY OUTCOMES:
HOAs | three months
  high order aberrations such as coma
Strehl Ratio | three months
  The derivative of point spread function (PSF)
objective visual quality | three months
  The modulation transfer function (MTF) curve
contrast sensitivity | three months
  Contrast sensitivity were obtained from the Functional Vision Analyzer
visual functions | three months
  Visual functions were obtained from the OCULUS Binoptometer 4P
IOL condition | three months
  IOL condition were obtained from the wavefront mode of the OPD-Scan III aberrometer.
subjective satisfaction | three years
  Satisfaction Questionnaire
photic phenomena | three years
  Questionnaire of photic phenomena

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Study Director — Department of Ophthalmology, Eye and Ear, Nose, and Throat Hospital, Fudan University

IPD SHARING:
Plan to Share IPD: Undecided